CLINICAL TRIAL: NCT03719118
Title: Effectiveness of Tailored Therapeutic Model According to the Expression of Genes Related to Immunomodulator-induced Myelosuppression in Inflammatory Bowel Disease Patients
Brief Title: Tailored Therapeutic Model According to the Expression of Genes in Inflammatory Bowel Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2015-0812
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotyping group (Experimental): The patients undergo pretreatment of genotyping for three genes (TPMT, NUDT15 and FTO)
  Interventions: Genetic: genotyping for three genes (TPMT, NUDT15 and FTO)
- Non-genotyping group (Active Comparator): Patients receive standard doses of thiopurines based on the conventional regimen without pretreatment genotyping.
  Interventions: Other: non-genotyping

INTERVENTIONS:
Genetic: genotyping for three genes (TPMT, NUDT15 and FTO) — Patients who carry any heterozygotic variants receive 50 mg AZA or 25 mg 6-mercaptopurine (6-MP), while those who have any homozygotic variants are recommended to take other alternative drugs instead of thiopurines
  Arms: Genotyping group
Other: non-genotyping — Patients receive standard doses of thiopurines based on the conventional regimen without pretreatment genotyping. Conventional regimen starts with 50 mg of AZA, then the dose is increased by 25 mg in every 1-2 weeks to 2.0-2.5 mg/kg along with regular monitoring of general blood tests including WBC counts.
  Arms: Non-genotyping group

SUMMARY:
This study is a randomized controlled study conducted at five tertiary university hospitals. Patients who are 20-80 years old, diagnosed as having Inflammatory Bowel Disease(IBD) and who are planned to start thiopurines for the first time for the treatment of IBD are enrolled. Patients are assigned to the genotyping group or to the non-genotyping group. The patients who carry any heterozygotic variant among the three genes receive 50 mg azathioprine (AZA) or 25 mg of 6-mercaptopurine, while those who have any homozygotic variant are recommended to take other alternative drugs. The patients who do not carry any genetic variant or are assigned in non-genotyping group receive the standard dose of thiopurines based on the conventional approach.

Patients in the non-genotyping group receive the standard dose of thiopurines based on the conventional approach.

ELIGIBILITY:
Inclusion Criteria:

* 20-80 years old
* Patients who were diagnosed as having IBD based on clinical, endoscopic, radiographic, and histological assessments,
* Patients who were planned to start thiopurines for the first time for the treatment of IBD.

Exclusion Criteria:

* Patients who had previous use of thiopurine
* Those who had abnormal laboratory findings prior to screening, including white blood cell (WBC) count < 3,000/μL, platelet (PLT) count < 100/μL, or elevation of aminotransferase more than twice the upper normal limits
* Those who were diagnosed other infectious diseases at the time of screening or receiving antibiotics within the previous 7 days;
* Those who were pregnant or lactating.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of myelosuppression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hee Cheon, MD, Principal Investigator — Severance Hospital
Locations (5):
- South Korea (5):
  - Severance Hospital, Seoul
  - Ewha Medical Research Institute, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet.

REFERENCES:
- [Derived] Chang JY, Park SJ, Jung ES, Jung SA, Moon CM, Chun J, Park JJ, Kim ES, Park Y, Kim TI, Kim WH, Cheon JH. Genotype-based Treatment With Thiopurine Reduces Incidence of Myelosuppression in Patients With Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2020 Aug;18(9):2010-2018.e2. doi: 10.1016/j.cgh.2019.08.034. Epub 2019 Aug 22. PMID 31446180